CLINICAL TRIAL: NCT06657131
Title: Diagnostic Performance and Clinical Impact of [18F]PSMA-1007 in the Context of Biochemical Recurrence of Prostate Cancer: a Real-World Evidence from a Monocentric, Prospective Observational Phase-4-Trial
Brief Title: Diagnostic Performance of [18F]PSMA-1007 in the Context of Biochemical Recurrence of Prostate Cancer
Acronym: [18F]PSMA-1007
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Emil Novruzov, Board Certified Nuclear medicine Physician, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2024-2995
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer After a Radical Treatment; Biochemical Recurrence of Malignant Neoplasm of Prostate; Biochemical Persistence of Prostate Cancer
Keywords: prostate cancer; biochemical recurrence; 18F-PSMA-1007; [18F]PSMA-1007; biochemical persistence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Following numerous retrospective studies and Phase-3-Studies with promising results, [18F]PSMA-1007 has been approved by european authorities. Therefore, it is a growing deployment of this diagnostic method anticipated. This study aims to investigate the diagnostic performance and clinical impact in a real-world-evidence in the context of regular clinical care. The evidence generated by this approach is supposed to assist in optimizing the management of prostate cancer patients.

DETAILED DESCRIPTION:
The advent of PSMA diagnostics and therapy has constituted a paradigm shift in the management of prostate cancer, supplanting other clinical and radiological diagnostic techniques. Consequently, [18F]PSMA-1007 (Radelumin®) has been approved in several EU countries, most recently in Germany in 2024, for use in primary staging of high-risk prostate cancer and re-staging in the context of biochemical recurrence (BCR). This may be regarded as a landmark in the management of prostate cancer, with the potential to markedly enhance the uptake of PSMA-PET diagnostics in the coming years.

The intention is to generate evidence-based data in everyday clinical practice with this so-called Real-World-Evidence (RWE) study. The planned study will facilitate a more detailed analysis of the diagnostic accuracy of Radelumin® in everyday clinical practice. This will involve dedicated examinations of certain subgroups and the prospective generation of a complete, high-quality database for future use of artificial intelligence (AI).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Conduct of [18F]PSMA-1007 PET Imaging in the context of regular clinical care

Exclusion Criteria:

* Technical Flaws in the acquisition protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study investigates the diagnosic potential of PSMA-PET imaging in patients with a histopathologically proven prostate cancer. Therefore, all participants will be only biologically male patients.
Study Population: The patient cohort will consist of biologically male patients with a histopathologically proven prostate cancer following a curative-intent cancer therapy. These patients will be referred to our center due to suspected recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
PSA-Stratified Detection rate of [18F]PSMA-1007 in BCR | From the timepoint of recruitment on for a time frame of 6 months for each individual
  Assessment of detection rate of molecular imaging in accordance with composite reference method or histopathological validation, if available
Clinical Impact | From the timepoint of recruitment on for a time frame of 6 months for each individual
  The assesment of the anticipated rate of therapy change based on the PSMA-PET imaging for the patients with BCR

SECONDARY OUTCOMES:
Prognostic value of [18F]PSMA-1007 for the patients with BCR | From the timepoint of recruitment on for a time frame of 24 months for each individual
  Assessment of prognostic value of [18F]PSMA-1007 imaging in terms of recurrence-free Survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Lars Giesel, Prof. Dr., Medical Doctor, Study Chair — Department of Nuclear Medicine, Medical Faculty and University Hospital Duesseldorf, Heinrich-Heine-University Duesseldorf
Locations (1):
- Department of Nuclear Medicine, Medical Faculty and University Hospital Duesseldorf, Heinrich-Heine-University Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to provide the IPD including the patient characteristics and study protocol. On a reasonable request, the investigators would also provide patient data with respect to evaluation of primary and secondary outcomes.
Supporting Information: Study Protocol, ICF
Time Frame: From the completion of the first study year by December 2025 up to the study end.
Access Criteria: The investigators plan to operate according to official requests via E-mail or website of clinicaltrials.gov.

REFERENCES:
- [Background] Panagiotidis E, Fragkiadaki V, Papathanasiou N, Kypraios C, Liatsikos E, Klampatsas A, Paschali A, Exarhos D, Zarokosta F, Chatzipavlidou V, Apostolopoulos D, Datseris I. Comparison of 18F-PSMA-1007 and 18F-Choline PET/CT in prostate cancer patients with biochemical recurrence: a phase 3, prospective, multicenter, randomized study. Nucl Med Commun. 2023 Dec 1;44(12):1126-1134. doi: 10.1097/MNM.0000000000001770. Epub 2023 Oct 2. PMID 37779440
- [Background] Giesel FL, Will L, Kesch C, Freitag M, Kremer C, Merkle J, Neels OC, Cardinale J, Hadaschik B, Hohenfellner M, Kopka K, Haberkorn U, Kratochwil C. Biochemical Recurrence of Prostate Cancer: Initial Results with [18F]PSMA-1007 PET/CT. J Nucl Med. 2018 Apr;59(4):632-635. doi: 10.2967/jnumed.117.196329. Epub 2018 Feb 1. PMID 29419475
- [Background] Cardinale J, Schafer M, Benesova M, Bauder-Wust U, Leotta K, Eder M, Neels OC, Haberkorn U, Giesel FL, Kopka K. Preclinical Evaluation of 18F-PSMA-1007, a New Prostate-Specific Membrane Antigen Ligand for Prostate Cancer Imaging. J Nucl Med. 2017 Mar;58(3):425-431. doi: 10.2967/jnumed.116.181768. Epub 2016 Oct 27. PMID 27789722